CLINICAL TRIAL: NCT02733523
Title: Promoting Self-Management, Health Literacy And Social Capital In Socioeconomically Disadvantaged Older Adults To Reduce Later Life Health Inequalities: A Randomized Clinical Trial
Brief Title: Self-management, Health Literacy and Social Capital in Socioeconomically Disadvantaged Older Adults
Acronym: AEQUALIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio Salut i Envelliment UAB (Other)
Collaborators: Recercaixa (Unknown); Equip Atencio Primaria Sardenya (Unknown)
Responsible Party: Principal Investigator, Laura Coll, MD, head of research on health and ageing, Fundacio Salut i Envelliment UAB
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FSIE-Recercaixa2014
Record Dates: First submitted 2016-02-10; First posted 2016-04-11 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Health Status Disparities; Subjective Health; Self Care; Social Capital; Health Literacy; Aging

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Program "Sentirnos bien" (Experimental): The intervention Program "Sentirnos bien" is based around a group dynamic, held once a week during 3 months, aimed at:
  1. Promoting the uptake of self-care healthy habits
  2. Promoting social capital at individual level:
  3. Promoting health literacy
  Interventions: Behavioral: Program "Sentirnos bien" (Feeling well)
- Control arm (No Intervention): The control arm will receive no intervention. Once the trial is finished, i.e. after the last follow-up evaluation, this arm will receive the intervention (waiting-list approach).

INTERVENTIONS:
Behavioral: Program "Sentirnos bien" (Feeling well) — Group-based intervention delivered face-to face and held once a week during 3 months. It comprises:
  1. Promoting the uptake of self-care healthy habits: providing information, setting personal goals and sharing experiences to facilitate behavioural change, specially on physical activity and healthy dietary habits.
  2. Promoting social capital at individual level: facilitating mutual knowledge and mutual support among participants and fostering participation in sociocultural and community activities in the neighbourhood through visits to the community assets accompanied by volunteers.
  3. Promoting health literacy: improving navigation through the health care system, communication with health professionals, as well as the understanding and decision making when buying food.
  Arms: Program "Sentirnos bien"

SUMMARY:
Motivations:

Socio-economic and education determinants have a big impact on health outcomes, in terms of worse health status in populations living in more disadvantaged conditions. Social capital, self-management and health literacy are some of the intermediate determinants, with the potential to mitigate health inequalities through interventions driven by local health agents. These three determinants are intensely interlinked and have, separately, impacts on self-perceived health. Social capital is defined in this project as an umbrella concept, which includes quantitative aspects of social resources (structural social capital: social networks and contacts, social and civic participation) as well as qualitative or subjective aspects (cognitive social capital: perceived social support, feeling of belonging and trust) and covers relations between subjects at a micro or individual level (family and friends) as well as at a macro or community level. Health literacy is understood as cognitive and social skills which determine the motivation and ability of individuals to gain access to, understand and use information in ways which promote and maintain good health. Both are key aspects for self-management behaviours. The target of our research project are older people living in urban socioeconomically disadvantaged areas, since ageing is in itself an inequality axis and urban environments concentrate the highest health disparities.

Objectives: With the aim to reduce health inequality, an intervention has been designed to promote self-management, health literacy and social capital among older people who perceived their health as fair or poor and are living in urban socioeconomically disadvantaged areas with the aim of improving their self-perceived health. Secondarily, the efficacy of the intervention will be analysed in terms of increasing self-management, health literacy and social capital (social support and social participation), quality of life, mental health and healthy lifestyles.

In third place, behavioural health patterns will be identified in relation to health literacy, social capital, gender, socioeconomic and educational level, and they will be linked to the intervention efficacy levels.

ELIGIBILITY:
Inclusion Criteria:

* community-dwelling older adults living in the urban areas of Barcelona, Blanes or Reus in socio-economically disadvantaged neighbourhoods.
* perception of their health as regular or bad according to the first question of the 12 items Short Form Survey from the RAND Medical Outcomes Study.

Exclusion Criteria:

* dependency to go to the local primary care center
* cognitive decline or dementia as diagnose
* any health condition that contraindicates physical activity
* terminal illness
* severe mental health disorders that difficult participating in a group dynamic

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Self-perceived health | at 3 months (just after the intervention)
  Same question than the 12 items Short Form Survey from the RAND Medical Outcomes Study. Answers will be recategorized as positive perception (excellent, very good or good) vs negative (regular or bad)

SECONDARY OUTCOMES:
Self-perceived health | at month 3 (just after the intervention) and at month 12 (9 months after the intervention)
  Thermometer from 0-100
Health related quality of life | at month 3 (just after the intervention) and at month 12 (9 months after the intervention)
  12 items Short Form Survey from the RAND Medical Outcomes Study.
Self-rated quality of life | t month 3 (just after the intervention) and at month 12 (9 months after the intervention)
  Thermometer from 0-100
Loneliness | t month 3 (just after the intervention) and at month 12 (9 months after the intervention)
  Scale Gierveld and De Jong
Depressive symptoms | at month 3 (just after the intervention) and at month 12 (9 months after the intervention)
  Geriatric Depression Scale
Physical activity | at month 3 (just after the intervention) and at month 12 (9 months after the intervention)
  International Physical Activity Questionnaire (IPAQ)
Short Physical Performance Battery | at month 3 (just after the intervention) and at month 12 (9 months after the intervention)
  Functional test that scores performance in three physical aspects: balance, strength and gait speed.
Health service use | at month 3 (just after the intervention) and at month 12 (9 months after the intervention)
  Times attending primary and hospital health care
Unintended effects | at month 3 (just after the intervention) and at month 12 (9 months after the intervention)
  Questions ad hoc to assess effects not intended by the intervention perceived negatively by the participant.
Self-care / healthy habits | at month 3 (just after the intervention) and at month 12 (9 months after the intervention)
  Scale ASA (Appraisal of Self-Care Agency Scale)
Health literacy | at month 3 (just after the intervention) and at month 12 (9 months after the intervention)
  questions from the European Health Literacy Scale (HLS EU-16)
Social capital | at month 3 (just after the intervention) and at month 12 (9 months after the intervention)
  2 questions from the European Values Survey
Social support | at month 3 (just after the intervention) and at month 12 (9 months after the intervention)
  Questionnaire "Inventario de recursos sociales en ancianos" from Díaz Veiga
Social participation | at month 3 (just after the intervention) and at month 12 (9 months after the intervention)
  Questionnaire "Escala Este II de Soledad - Índice de participación social subjetiva"

CONTACTS AND LOCATIONS:
Overall Officials: Laura Coll-Planas, MD, Principal Investigator — Fundació Salut i Envelliment UAB; Sergi Blancafort, PhD, Principal Investigator — Fundació Salut i Envelliment UAB; Rosa Monteserin, MD PhD, Principal Investigator — Equipo Atencio Primaria Sardenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berkman ND, Sheridan SL, Donahue KE, Halpern DJ, Crotty K. Low health literacy and health outcomes: an updated systematic review. Ann Intern Med. 2011 Jul 19;155(2):97-107. doi: 10.7326/0003-4819-155-2-201107190-00005. PMID 21768583
- [Background] Foster G, Taylor SJ, Eldridge SE, Ramsay J, Griffiths CJ. Self-management education programmes by lay leaders for people with chronic conditions. Cochrane Database Syst Rev. 2007 Oct 17;(4):CD005108. doi: 10.1002/14651858.CD005108.pub2. PMID 17943839
- [Background] Fried LP, Carlson MC, Freedman M, Frick KD, Glass TA, Hill J, McGill S, Rebok GW, Seeman T, Tielsch J, Wasik BA, Zeger S. A social model for health promotion for an aging population: initial evidence on the Experience Corps model. J Urban Health. 2004 Mar;81(1):64-78. doi: 10.1093/jurban/jth094. PMID 15047786
- [Background] Ahnquist J, Wamala SP, Lindstrom M. Social determinants of health--a question of social or economic capital? Interaction effects of socioeconomic factors on health outcomes. Soc Sci Med. 2012 Mar;74(6):930-9. doi: 10.1016/j.socscimed.2011.11.026. Epub 2012 Jan 21. PMID 22305807
- [Background] Kawachi I, Kennedy BP, Glass R. Social capital and self-rated health: a contextual analysis. Am J Public Health. 1999 Aug;89(8):1187-93. doi: 10.2105/ajph.89.8.1187. PMID 10432904
- [Background] Nyqvist F, Forsman AK, Giuntoli G, Cattan M. Social capital as a resource for mental well-being in older people: a systematic review. Aging Ment Health. 2013;17(4):394-410. doi: 10.1080/13607863.2012.742490. Epub 2012 Nov 27. PMID 23186534
- [Derived] Blancafort Alias S, Monteserin Nadal R, Moral I, Roque Figols M, Rojano I Luque X, Coll-Planas L. Promoting social capital, self-management and health literacy in older adults through a group-based intervention delivered in low-income urban areas: results of the randomized trial AEQUALIS. BMC Public Health. 2021 Jan 7;21(1):84. doi: 10.1186/s12889-020-10094-9. PMID 33413233
- [Derived] Coll-Planas L, Blancafort S, Rojano X, Roque M, Monteserin R. Promoting self-management, health literacy and social capital to reduce health inequalities in older adults living in urban disadvantaged areas: protocol of the randomised controlled trial AEQUALIS. BMC Public Health. 2018 Mar 13;18(1):345. doi: 10.1186/s12889-018-5219-x. PMID 29534699